CLINICAL TRIAL: NCT05524961
Title: Randomized Placebo- and Active-controlled Trial for Assessing the Efficacy of Bright Light Therapy for Sleep and Mood Symptoms in Patients With Parkinson's Disease
Brief Title: Bright Light Therapy for Non-motor Symptoms in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Joey WY Chan, Clinical Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021.676T
Record Dates: First submitted 2022-08-25; First posted 2022-09-01 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Light therapy; Daytime sleepiness; Non-motor symptom
MeSH Terms: conditions — Parkinson Disease; Disorders of Excessive Somnolence | interventions — Ultraviolet Therapy

STUDY DESIGN:
Intervention Model Description: Randomized placebo- and active-controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The subjects will be explained that the study aims to test the efficacy of the different modalities of non-pharmacological treatments for depression including bright light therapy and the negative ion generator, without mentioning which one is the placebo. An independent outcome assessor will be blinded to the treatment allocation throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Timed-Bright light therapy (BLT group) (Experimental): 10,000lux bright light
  Interventions: Device: Bright light therapy
- Timed-inactivated negative ion generator (Active-control group) (Active Comparator): Inactivated negative ion generator
  Interventions: Device: Inactivated negative ion generator
- Random-time inactivated negative ion generator (placebo group) (Placebo Comparator): Inactivated negative ion generator
  Interventions: Device: Inactivated negative ion generator

INTERVENTIONS:
Device: Bright light therapy — Regularly-timed exposure to 10,000lux bright light therapy for 60minutes a day for six weeks
  Arms: Timed-Bright light therapy (BLT group)
Device: Inactivated negative ion generator — Regularly-timed exposure to an inactivated negative ion generator for 60minutes a day for six weeks
  Arms: Timed-inactivated negative ion generator (Active-control group)
Device: Inactivated negative ion generator — Randomly-timed exposure to an inactivated negative ion generator for 60minutes a day for six weeks
  Arms: Random-time inactivated negative ion generator (placebo group)

SUMMARY:
This is a randomized placebo- and active-controlled trial for assessing the efficacy of bright light therapy for sleep and mood symptoms in patients with Parkinson's disease

DETAILED DESCRIPTION:
The primary aim of this study is to compare the efficacy of timed-BLT (BLT group) in reducing excessive daytime sleepiness in patients with Parkinson's disease, when compared to a timed-inactivated negative ion generator (active-control group).

The secondary aims of the study are to examine the effect of timed-BLT on other non-motor symptoms, including depression, fatigue; and the quality of life.

Additional analyses will be carried out to examine the efficacy of the timed-placebo as compared to the random-time placebo (placebo group).

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic Parkinson's disease diagnosed by neurologist according to the UK Parkinson's Disease Society Brain Bank clinical diagnostic criteria
2. Capable to give informed consent
3. Maintained on stable dose of medications for Parkinson's disease/psychotropic drugs for at least four weeks prior to entry of the study
4. Score 14 or more on the Epworth Sleepiness Scale

Exclusion Criteria:

1. A current or past history of manic or hypomanic episode, schizophrenia, mental retardation, or substance use disorder. (Subjects with depression or anxiety disorders will not be excluded)
2. Unstable medical or psychiatric condition
3. Presence of substantial suicidal risk as judged by the clinician and/or screening instruments
4. Presence of active psychotic symptoms that might impair the ability to consent or validity of the interview
5. Cognitive impairment with score of 19 or below by the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA)
6. Contraindication to bright light therapy: history of light induced migraine. Epilepsy, current use of photosensitizing medications, presence of eye disease, e.g. retinal disease, severe cataract, glaucoma and blindness
7. Significant medical condition/ hearing impairment/ speech deficit lead to incapability in completing clinical interview
8. Regular shift worker or trans-meridian flight in the past three months
9. Enrolment in another clinical trial of an investigational medicinal product or device
10. Subjects who are on exogenous melatonin
11. Patients with deep brain stimulation (DBS) implant
12. Patients with known sleep disorders, eg. untreated severe sleep apnea, restless leg syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of daytime sleepiness | at the end of 6-week treatment
  Change in the score of Epworth Sleepiness Scale (ESS), ESS score ranges from 0-24, higher score indicates greater sleepiness

SECONDARY OUTCOMES:
Change of depressive symptoms | at the end of 6-week treatment
  Change in the score of Montgomery-Åsberg Depression Rating Scale (MADRS), MARDS ranges from 0-60, higher score indicates greater severity of depressive symptoms
Change in fatigue symptoms | at the end of 6-week treatment
  Change in the score of Faitgue Severity Scale (FSS), FSS consists of 9 items and each as rated on a scale from 1-7, higher score indicates greater severity of fatigue
Change in quality of life | at the end of 6-week treatment
  Change in score of Short-Form 12-item (SF-12) scale. SF-12 consists of two subscales - a mental component score (MCS-12) and a physical component score (PCS-12), a higher score indicates better quality of life. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No